CLINICAL TRIAL: NCT07023263
Title: Evaluation of Perioperative Anesthesia Effectiveness in Hysteroscopy Cases Administered With Target-Controlled Infusion (TCI)
Brief Title: Target-Controlled Infusion (TCI) Effectiveness in Hysteroscopy
Status: Active, not recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Demet Coşkun, Prof., Gazi University
Other Study IDs: 2024-KAEK-07
Record Dates: First submitted 2025-05-19; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia Depth Monitoring; Analgesia Assessment; Perioperative Safety and Recovery; Target Controlled İnfusion
Keywords: Hysteroscopy; Target-Controlled Infusion (TCI); Eleveld; Schnider; Minto; Consciousness Monitoring; Anesthetic Depth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Standart TCI model group: Patients in this group will receive general anesthesia using Target-Controlled Infusion (TCI) with the Schnider model for propofol and the Minto model for remifentanil.
  Interventions: Device: Schnider+ Mİnto
- Eleveld TCI Model Group: Patients in this group will receive general anesthesia using the Eleveld model for both propofol and remifentanil
  Interventions: Device: Eleveld

INTERVENTIONS:
Device: Schnider+ Mİnto — Patients assigned to the Standart TCI model Group would have Schnider + Minto models throughout the surgery. The patients would be monitorized with anesthesia depth, analgesia monitoring, NIRS, and recovery parameters.
  Groups: Standart TCI model group
Device: Eleveld — Patients assigned to the Eleveld TCI model Group would have Eleveld+Eleveld models throughout the surgery. The patients would be monitorized with anesthesia depth, analgesia monitoring, NIRS, and recovery parameters.
  Groups: Eleveld TCI Model Group

SUMMARY:
This prospective, randomized, observational study aims to evaluate the perioperative anesthetic efficacy of different Target-Controlled Infusion (TCI) models-specifically Minto, Schnider, and Eleveld pharmacokinetic models-in patients undergoing hysteroscopy under general anesthesia. 90 female patients will be randomized into two groups, each receiving different TCI model combinations for propofol and remifentanil. Primary outcomes include intraoperative consciousness (BIS/SEF), analgesia (ANI), tissue oxygenation (NIRS), and recovery parameters. The study seeks to identify model-specific benefits regarding patient and surgeon satisfaction, recovery time, and complication rates.

DETAILED DESCRIPTION:
This study aims to evaluate the perioperative anesthetic efficacy of target-controlled infusion (TCI) in hysteroscopy cases. The study will be conducted in the Gynecology and Obstetrics Operating Room located on the 9th floor of Gazi University Hospital between April 2025 and July 2025.

The study will include women aged 18-65 years who will undergo hysteroscopy and meet the criteria of ASA I-II classification, with no significant comorbidities and a BMI < 35. The study is planned in two groups, with each group consisting of 45 patients, totaling 90 participants.

In the first group, TCI protocols based on the Schnider and Minto models will be applied. The initial target concentrations for propofol and remifentanil infusion will be set at 5 µg/mL and 4 ng/mL, respectively. In the second group, the Eleveld model will be used. The propofol dose will be adjusted according to the patient's age using the Eleveld algorithm, and the remifentanil effect-site concentration will be maintained at 3 ng/mL.

Participants will be informed about the study, and those eligible and willing to participate will provide signed informed consent. Upon being brought to the operating room, intravenous access will be checked and established if not already in place. Non-invasive blood pressure, heart rate, and oxygen saturation will be monitored in accordance with ASA standards.

Following this, Masimo Root device with SedLine, NIRS, and ANI sensors will be attached to the appropriate sites on the patients, ensuring data flow. These sensors will continuously monitor the patient's level of consciousness, tissue oxygenation, and pain response.

The Braun Space Plus Perfusor will be utilized as the TCI device. Patient-specific data, including age, height, weight, and gender, will be entered, and the effect-site concentrations for propofol and remifentanil will be set according to the respective TCI model being applied. Once all settings are confirmed and the device is operational, TCI infusion will be initiated.

After achieving loss of consciousness, a Laryngeal Mask Airway (LMA) of appropriate size will be inserted, and the patient will be connected to a ventilator. During the procedure, TCI infusion rates will be adjusted to maintain a SedLine value between 25-50 for propofol and an ANI range of 50-70 for remifentanil, ensuring hemodynamic stability.

Throughout the operation, hemodynamic data, SedLine, NIRS, and ANI values will be continuously monitored and recorded at specified intervals in the Case Report Form (CRF). The concentrations and total amounts of propofol and remifentanil administered will also be regularly monitored and documented.

Upon completion of the surgical procedure and initiation of hemostasis, TCI infusion will be terminated. Patients with increased SedLine values will have their LMAs removed when appropriate, and those who are alert and without respiratory distress will be transferred to the recovery room. In this phase, hemodynamic parameters, VAS pain scores, Aldrete scores, and nausea/vomiting status will be assessed and recorded. Patients achieving an Aldrete score of 10, who are hemodynamically stable and without complications, will be transferred to the service ward.

Additionally, patient and surgeon satisfaction will be evaluated and recorded in the CRF. All data will be analyzed using SPSS 27.0 software. Intraoperative drug consumption, time to loss of consciousness, recovery duration, and complication rates will be analyzed using ANOVA. Correlation analyses will assess the relationships between drug consumption and recovery times.

Confidentiality will be strictly maintained throughout the study. Data will be accessible only to the research team and will be coded to ensure participant anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-65
* ASA I-II
* Scheduled for hysteroscopy under general anesthesia
* Signed informed consent

Exclusion Criteria:

* Allergy to study drugs
* Significant cardiac, pulmonary, neurological disease
* Pregnancy or breastfeeding
* BMI >35
* Substance use disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include female patients aged 18 to 65 years who are scheduled to undergo elective hysteroscopic surgery under general anesthesia. Eligible participants must be classified as ASA Physical Status I-II, with no significant comorbidities. All patients will provide written informed consent prior to enrollment.
  Patients with a history of significant cardiac, pulmonary, or neurological disease, known allergies to propofol or remifentanil, pregnancy or breastfeeding status, body mass index (BMI) >35, or substance use disorder will be excluded.
  A total of 90 patients will be randomized into two groups (45 patients each) to receive anesthesia with different TCI models. The study population is limited to a single academic tertiary care center (Gazi University Faculty of Medicine, Department of Anesthesiology and Reanimation).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intraoperative Complications | perioperative period: from beginning of anesthesia induction to discharge from recovery room
  Number of patients experiencing at least one predefined complication during anesthesia, including hypotension (MAP <65 mmHg >1 min), bradycardia (HR <50 bpm), or oxygen desaturation (SpO₂ <92%)
Total Recovery Time Until Discharge Readiness | Up to 2 hours post-anesthesia
  Time elapsed from cessation of anesthetic agents to achieving an Aldrete score ≥9

SECONDARY OUTCOMES:
Total Propofol Consumption | From induction to end of anesthesia
  Total amount of propofol (mg) administered via TCI during the entire anesthetic period
Total Remifentanil Consumption | From induction to end of anesthesia
  Total amount of remifentanil (mcg) administered via TCI during the entire anesthetic period
Patient and Surgeon Satisfaction and Willingness to Repeat the Same Anesthesia Method | Patient: Within 1 hour postoperatively (before recovery room discharge) Surgeon: Immediately after surgery
  The percentage of cases in which both the patient and the operating surgeon answered "Yes" to the question:
  Patient: "Would you prefer the same anesthesia technique again in the future?" Surgeon: "Would you prefer the same anesthetic method for future similar cases?"
Incidence of Postoperative Nausea and Vomiting (PONV) | Within 2 hours after anesthesia discontinuation
  Number of patients who experience at least one episode of nausea and/or vomiting during the early recovery period
Incidence of Postoperative Pain | Within 30 minutes after arrival in the recovery room
  Number of patients reporting a pain score ≥4 on a 0-10 Numerical Rating Scale (NRS) during recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol